CLINICAL TRIAL: NCT02174341
Title: Investigate the Prevalence of Serum Chikungunya Virus Infection, and Against Those Suspected Dengue Fever, Chikungunya Disease-related Tests Conducted
Brief Title: The Pilot Study of Chikungunya Virus Infections in Southern Taiwan
Status: Completed | Type: Observational
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KMUH-IRB-20110428
Record Dates: First submitted 2014-06-20; First posted 2014-06-25 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Chikungunya Fever
Keywords: Chikungunya fever; Chikungunya Virus
MeSH Terms: conditions — Chikungunya Fever

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This test is to be collected during the dengue outbreak samples, including samples back in the past and forward to close the case, investigating the prevalence of serum Chikungunya virus infection, and against those suspected dengue fever, Chikungunya disease-related tests conducted to clarify dengue and Chikungunya disease of clinical judgment, rapid method to detect Chikungunya virus and then develop.

DETAILED DESCRIPTION:
During the execution of this project was ended March 1, 2012 to December 31, 2015, is expected to gather 300 suspected dengue infection, of whom 150 dengue-negative test results, test results of 150 dengue positive. And closed the case into prospective and retrospective analysis of the last sample into two parts.

Case closed after part of a prospective analysis of the study, subjects were required to complete consent forms and collect 20 ml blood samples, blood samples will be checked to identify dengue and Chikungunya disease associated serum antigen-antibody reaction , PCR (polymerase chain reaction) test and sequence analysis and pathogen identification and separation, in order to identify the source of infection difference. In addition, retrospective analysis of the last part of the specimen, sucked "after the health of the host track dengue infection, host immune regulation changes, and possible interactions with viral hepatitis" (KMUH-IRB-960195) collected by the inspection plan body, the number of samples included in the plan to close the case, and contact with the subjects, changes to inform the content of the plan to re-sign the consent form.

ELIGIBILITY:
Inclusion Criteria:

* Suspected of being infected with dengue fever

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The samples are obtained from the Kaohsiung Medical University Chung-Ho Memorial Hospital in Kaohsiung, Taiwan.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2012-04; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
For persons with suspected dengue fever, Chikungunya disease-related testing conducted to clarify the clinical dengue and Chikungunya disease of judgment | 75 months
  The project expects to help physicians understand overview of Taiwan Chikungunya epidemic diseases and assisting their clinical judgment. Hope to establish a complete ilk disease and clinical information, and then establish a rapid detection of Chikungunya virus.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaoshing Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan